CLINICAL TRIAL: NCT00832624
Title: Open-label, Non Placebo-Controlled Study To Verify the Effect of Sitagliptin In Adult Patients With Type 2 Diabetes and Inadequate Glycemic Control
Brief Title: The Effect of Sitagliptin in Type 2 Diabetes Mellitus With Inadequate Glycemic Control (MK0431-118)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0431-118; 2009_526
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Results first posted 2010-10-11 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus Non-insulin-dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): sitagliptin
  Interventions: Drug: sitagliptin

INTERVENTIONS:
Drug: sitagliptin — Sitagliptin, 100 mg, 1 Tablet, once a day, for 18 weeks
  Other Names: Januvia; MK0431

SUMMARY:
to assess the effect of treatment with Sitagliptin (MK0431) on HbA1c (Hemoglobin A1c) and the safety and tolerability of Sitagliptin.

ELIGIBILITY:
Inclusion Criteria:

* Patients Who Are 18 Years Of Age With Type 2 Diabetes Mellitus Who Are Either:

  * Not On Antihyperglycemic (AHa) Medication (Off For At Least 2 Months)
  * Or On A Single AHa

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-11-26 (Actual); Primary Completion 2009-09-02 (Actual); Study Completion 2009-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment process occurred in the Hospital Regional de Taguatinga between November, 26 2008 and May, 27 2009.
  First Patient in: 26-Nov-2008; Last patient in: 27- May- 2009
Pre-assignment Details: Patients between 18 and 75 years old with type 2 diabetes mellitus (T2DM) and inadequate glycemic control, who had not taken medication for at least 2 months or using a single drug for diabetes mellitus were enrolled in the study. Insulin-dependent patients were excluded from the study.
Groups:
- Sitagliptin 100 mg: Sitagliptin, 100 mg, 1 Tablet, once a day, for 18 weeks
Period: Overall Study
Arm/Group | Sitagliptin 100 mg
Started | 10
Completed | 0
Not Completed | 10
Not completed — Study Terminated | 10

BASELINE CHARACTERISTICS:
Arm/Group | Sitagliptin 100 mg
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Region of Enrollment [Number; unit: participants]
  Brazil | 10
Weight [Mean (Standard Deviation); unit: Kilograms] | 71.59 (11.55)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Hemoglobin A1c) at Week 18
Description: Glycosylated hemoglobin (HbA1c) was to be measured as the percentage of hemoglobin that has glucose bound to it; however, the study was terminated early therefore no laboratory tests were performed, and no outcome data was collected.
Time Frame: Baseline and Week 18
Population: The study was terminated early and no data were analyzed for this outcome.
Arm/Group | Sitagliptin 100 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The planned 18-week study was terminated early due to reconsideration of the study design.
Description: None of the 10 patients progressed beyond the second study visit, no laboratory tests were performed, and adverse experience data were not collected.
Arm/Group | Sitagliptin 100 mg
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The planned 18-week study was terminated early due to reconsideration of the study design. None of the 10 patients progressed beyond the second study visit, no laboratory tests were performed, and adverse experience data were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.